CLINICAL TRIAL: NCT05815420
Title: Home Tele-Monitoring of Non-Invasive Ventilation in Chronic Obstructive Pulmonary Disease in France
Brief Title: Home Tele-Monitoring of Non-Invasive Ventilation in COPD Patients in France
Acronym: HOV-C
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Association Nationale pour les Traitements A Domicile, les Innovations et la Recherche (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-A00565-40
Record Dates: First submitted 2023-04-04; First posted 2023-04-18 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Non invasive ventilation; Telemonitoring
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Noninvasive Ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Non invasive ventilation — Treatment by non invasive ventilation

SUMMARY:
Tele-monitoring emerged and unfolded differently among various healthcare organisations and countries. Evidence regarding its impact on the management of COPD patients is still insufficient to draw firm conclusions. Assumption has been made that remote monitoring of home NIV treatment could help to identify novel predictors of the early detection of NIV failure and deteriorations in patients with COPD.

The incidence in routine clinical care of unplanned all-cause and COPD-caused hospitalisations in patients treated with NIV therapy who are continuously monitored by telemetric data in France needs evaluation.

In addition, predictors of unplanned all-cause and COPD-caused hospitalisations as well as of compliance and persistence to NIV therapy should be assessed in this patient population with special respect to continuous tele-monitoring.

The study will determine in France the incidence in routine clinical care of unplanned all-cause and COPD-caused hospitalisations in patients treated with NIV therapy who are continuously monitored by telemetric data. Clinical and telemetric predictors of unplanned all-cause and COPD-caused hospitalisations and of NIV therapy compliance and persistence will be assessed in those patients

ELIGIBILITY:
Inclusion criteria:

* Age ≥18 years
* COPD eligible for NIV treatment
* Prescription of an adequate ResMed NIV device with tele-monitoring option as part of routine clinical care
* Acceptance of tele-monitoring and corresponding data handling
* Naive to long-term NIV treatment with initiation of NIV either ≤7 days before or after enrolment into study
* Able to fully understand information on data protection and provide written informed consent for use of corresponding medical and telemetric data.

Exclusion criteria:

* Invasive ventilation therapy
* Another life-threatening disease with estimated survival < 12 months (other than COPD, e.g. cancer)
* Further exclusion criteria according to manua of the device intended and prescribed

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD Patient with a first prescription of NIV treatment
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of unplanned all-cause hospitalisations in routine clinical care in patients treated with NIV therapy who are continuously monitored by telemetric data | 1 year
  Rate of unplanned all-cause hospitalisations in the study population normalised to one year of follow up